CLINICAL TRIAL: NCT01365325
Title: Management of Chronic Heart Failure: Role of the Handled Echocardiography in Home Monitoring Care Programs
Brief Title: Handled Echocardiography and Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Ugo Oliviero, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 228/08
Record Dates: First submitted 2011-05-27; First posted 2011-06-03 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2010-12

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — epicatechin gallate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- handled echocardiography (Experimental): home monitoring care program based on clinical and electrocardiographic evaluations and periodical handled echocardiographic examinations
  Interventions: Other: handled echocardiography in home monitoring program
- home monitoring program (Active Comparator): home monitoring care program based on clinical and electrocardiographic evaluations
  Interventions: Other: ecg and clinical evaluation in home monitoring program

INTERVENTIONS:
Other: handled echocardiography in home monitoring program — home monitoring with clinical evaluations and ECG every three months and echocardiography examinations at the 6th, 12th and 18th month
  Other Names: Handled echocardiography
  Arms: handled echocardiography
Other: ecg and clinical evaluation in home monitoring program — home monitoring with clinical evaluations and ECG every three months
  Other Names: home monitoring with clinical evaluations and ECG
  Arms: home monitoring program

SUMMARY:
The aim of the study is to compare two different home monitoring care programs in patients with chronic heart failure in functional class NYHA III, one of them based on clinical and electrocardiographic evaluations, the other one using also periodical handled echocardiographic examinations.

DETAILED DESCRIPTION:
Randomized, blinded, controlled, monocentric study comparing two different home monitoring care programs in patients with chronic heart failure in functional class NYHA III, one of them based on clinical and electrocardiographic evaluations every three months, the other one using also periodical handheld echocardiographic examinations at the 6th, 12th and 18th month.

The events occurring during the 18 month follow up and the results of the final echocardiography performed in all the patients will be transmitted to and evaluated by an independent observer, unaware of the features of the follow up. At the end of the trial, the randomization code will be opened and the events will be ascribed to the two groups. The primary end point is rehospitalization for worsening of heart failure symptoms and/or for the appearance of major vascular events during the 18 months follow up. Secondary end points include home treated vascular events, cardiovascular death and the composite end point death + rehospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Heart Failure in functional class NYHA III
* At least once hospitalization during the last year for worsening of clinical symptoms or for the appearance of acute cardiovascular events
* Patients who cannot easily reach the pertaining Sanitary District for different reasons (i.e. the presence of architectural barriers, the absence of a lift, a too great distance between home and Sanitary District without someone helping)
* age ≥ 70 years
* written informed consent

Exclusion Criteria:

* Patients who were waiting for cardiac surgery or patients who had undergone a cardiac operation within three months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Rehospitalization for worsening of heart failure symptoms and/or for the appearance of major vascular events | 18 months

SECONDARY OUTCOMES:
Home treated major vascular events | 18 months
  Number of Participants with major vascular events occurred during the 18 months follow up who did not go to the Hospital and were home treated
Cardiovascular death | 18 months
Composite end point death + rehospitalization | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Oliviero, MD, Principal Investigator — Federico II University
Locations (1):
- Federico II University, Naples, Italy